CLINICAL TRIAL: NCT00587951
Title: The Influence of SISCOM on Intracranial Electrode Implantation in Epilepsy Surgical Candidates
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. K. Meng Tan, Mayo Foundation
Other Study IDs: 2170-05
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-11

CONDITIONS: Epilepsy
Keywords: Clinical decision-making; Ictal SPECT; Epilepsy surgery
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Candidates for epilepsy surgery, undergoing pre-surgical evaluation at Mayo Clinic, and in whom SISCOM was ordered by the treating physician as part of that evaluation

SUMMARY:
The aim of this study is to determine the role of SISCOM (see below) in aiding clinicians to manage epilepsy surgery candidates. SISCOM is already a routine component of pre-surgical epilepsy evaluation at Mayo Clinic. In particular, we are interested in assessing whether use of SISCOM can minimize the need for prolonged (>24 hours) invasive monitoring with electrodes placed on the surface of the brain prior to surgical resection.

Note: this study has recruited the required number of patients and is closed to further enrolment.

DETAILED DESCRIPTION:
Successful epilepsy surgery depends on accurate identification of the area of brain from which seizures originate (the epileptogenic zone). There are many non-invasive tests (including EEG and MRI) to indicate this area. Some patients require implantation of intracranial electrodes in order to determine the epileptogenic zone. A test known as SISCOM (subtraction ictal-interictal SPECT co-registered with MRI) has been validated as a non-invasive means of indicating the epileptogenic zone. However, this test is not widely available in the US, and it is not known how often the additional information provided by SISCOM makes a difference to clinical decision-making.

In order to determine the contribution of SISCOM towards clinical decision-making in epilepsy surgery candidates, we will ask epileptologists at Mayo Clinic to consider case presentations given all clinical information except for SISCOM results, and then to reconsider those same cases in conjunction with SISCOM data. This will indicate the degree to which SISCOM influences decision making.

50 patients at Mayo Clinic (38 adults, 12 children) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of localization-related epilepsy
* Evaluated by clinical epileptologist at Mayo Clinic
* SISCOM ordered by treating physician
* Case presented at weekly Epilepsy Surgery Conference
* Patient consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients evaluated at Mayo Clinic and being considered for epilepsy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Category of management recommendation (proceed straight to surgical resection, intracranial electrode implantation, more imaging studies OR recommend medical rather than surgical management) | Instantaneous

CONTACTS AND LOCATIONS:
Overall Officials: Meng Tan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States